CLINICAL TRIAL: NCT00828373
Title: The Effect of Intravenous Lidocaine on the Time Course of Rocuronium Induced Neuromuscular Block. A Randomised, Placebo-controlled, Electrophysiological Study
Brief Title: The Influence of Intravenous Lidocaine on the Action of the Neuromuscular Blocker Rocuronium
Acronym: LidoRoc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Christoph Czarnetzki, MD, Division of Anesthesiology, University Hospitals of Geneva
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER 08 - 202; Swissmedic
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2009-08

CONDITIONS: Neuromuscular Block
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Placebo — Immediately before induction, patients will receive 0.15 ml kg-1 of the study drug as an intravenous bolus followed, after tracheal intubation, by a continuous intravenous infusion of 0.2 ml kg-1 h-1. In the Placebo group this will be physiologic saline. The infusion will be stopped after complete recovery from the neuromuscular block.
  Arms: Placebo
Drug: Lidocaine — Immediately before induction, patients will receive 0.15 ml kg-1 of the study drug as an intravenous bolus followed, after tracheal intubation, by a continuous intravenous infusion of 0.2 ml kg-1 h-1. In the lidocaine Arm this regimen corresponds to 1.5 mg kg-1 lidocaine bolus injection and 2 mg kg-1 h-1 lidocaine continuous infusion. The infusion will be stopped after complete recovery from the neuromuscular block.
  Other Names: Rapidocaïne®; Xylocain®
  Arms: Lidocaine

SUMMARY:
Lidocaine is a local anesthetic which is widely used in daily anesthesia and surgical practice. It has been shown that intravenous lidocaine given during an operation has analgesic properties. Finally intravenous lidocaine is inexpensive and easy to administer and safe if non-toxic doses are respected. It is likely that the use of lidocaine infusions during anesthesia might increase in the coming years. Neuromuscular blockers (curare like substances) are used in anesthesia to facilitate tracheal intubation and to achieve muscle relaxation and immobility during surgery. Rocuronium is one of the most widely used neuromuscular blocking agents. Local anesthetics, such as lidocaine, are known to potentiate the effect of neuromuscular blocking agents. In the study the investigators want to evaluate the effect of intravenous lidocaine during the operation on the time course of the rocuronium-induced neuromuscular block. A secondary aim is to evaluate intubation conditions (lidocaine has been shown also to improve intubation conditions) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age ≥18 to 60 years, male or female.
* American Society of Anesthesiology [ASA] status I or II.
* Patient is able to read and understand the information sheet and to sign and date the consent form.
* Patient scheduled of elective surgery lasting longer than 120 min without need for continuous curarisation.
* Surgery without application of local anesthetics (epidurals, wound-infiltration).
* If the patient is female and of childbearing potential, she must have a negative pregnancy test.

Exclusion Criteria:

* A history of allergy or hypersensitivity to rocuronium or lidocaine
* Neuromuscular disease
* Preoperative medications known to influence neuromuscular function (for instance, certain antibiotics [aminoglycosides] and anticonvulsants [phenytoine])
* Electrolyte abnormalities (for instance, hypermagnesemia)
* Hepatic or renal insufficiency
* Patients with epileptic disease
* Patients with a body mass index <19 or >28 kg m2
* Pregnant or breastfeeding women
* Expected difficult intubation or mask ventilation
* Atrioventricular heart block II or III -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Onset and recovery of the neuromuscular block | From start of injection of rocuronium until TOF 90%

SECONDARY OUTCOMES:
To evaluate intubation conditions at T1, we will use the scale according to the Good Clinical Research practice (GRCP) in neuromuscular research | 2 to 3 minutes
Any minor adverse event (no need for intervention) or major adverse event will be recorded. | up to 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Czarnetzki, MD, MBA, Principal Investigator — University Hospitals of Geneva; Martin R Tramèr, MD, Dphil, Study Chair — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Czarnetzki C, Lysakowski C, Elia N, Tramer MR. Intravenous lidocaine has no impact on rocuronium-induced neuromuscular block. Randomised study. Acta Anaesthesiol Scand. 2012 Apr;56(4):474-81. doi: 10.1111/j.1399-6576.2011.02625.x. Epub 2012 Jan 19. PMID 22260297